CLINICAL TRIAL: NCT04412707
Title: A Randomized, Two-period, Cross-over, Phase 2 Study, Comparing Pharmacokinetics, and Assessing Safety and Tolerability of Peripheral and Central i.v. Administration of Melphalan Flufenamide (Melflufen) in RRMM Patients
Brief Title: A PK, Safety and Tolerability Study of Peripheral and Central Infusion of Melflufen in RRMM Patients
Acronym: PORT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to terminate the study following an FDA request of a partial clinical hold.
Sponsor: Oncopeptides AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OP-109
Record Dates: First submitted 2020-05-18; First posted 2020-06-02 (Actual); Results first posted 2022-08-16 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-01

CONDITIONS: RRMM
Keywords: central intravenous administration; peripheral intravenous administration; central venous catheter (CVC); peripheral venous catheter (PVC)
MeSH Terms: interventions — Melphalan; melflufen; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Melflufen 40 mg iv Day 1 of each 28 day cycle. Dexamethasone 40 mg po Day 1,8, 15 and 22 of each 28 day cycle, if > 75 years of age 20 mg. Cycle 1 will be administered via a Peripheral Venous Catheter (PVC) and cycle 2 and onwards melflufen will be administered via a Central Venous Catheter (CVC).
  Interventions: Drug: Melphalan; Drug: Dexamethasone
- Arm B (Active Comparator): Melflufen 40 mg iv Day 1 of each 28 day cycle. Dexamethasone 40 mg po Day 1,8, 15 and 22 of each 28 day cycle, if > 75 years of age 20 mg. Cycle 1 will be administered via a Central Venous Catheter (CVC) and cycle 2 will be administered via a Peripheral Venous Catheter (PVC). From cycle 3 and onwards melflufen will be administered via CVC.
  Interventions: Drug: Melphalan; Drug: Dexamethasone

INTERVENTIONS:
Drug: Melphalan — Peripheral versus central administration
  Other Names: melflufen flufenamide
Drug: Dexamethasone — Oral tablets

SUMMARY:
This is a randomized, two-period, cross-over Phase 2 study, comparing PK, and assessing safety and tolerability and efficacy of peripheral and central intravenous administration of melflufen in patients with RRMM. It is an international study, enrolling patients in US and Europe. The study will enroll patients following at least 2 lines of prior therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or older
2. Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol;
3. A prior diagnosis of multiple myeloma (MM) with documented disease progression in need of treatment at time of screening;
4. Measurable disease defined as any of the following:

   * Serum monoclonal protein ≥ 0.5 g/dL by serum protein electrophoresis (SPEP)
   * ≥ 200 mg/24hr of monoclonal protein in the 24hour urine collection by electrophoresis (UPEP)
   * Serum free light chain (SFLC) ≥ 10 mg/dL AND abnormal serum kappa to lambda free light chain (FLC) ratio
5. Received at least 2 prior lines of therapy and is refractory to an immunomodulatory drug (IMiD) and a proteasome inhibitor (PI). The definition of refractory includes intolerance to an IMiD/PI after at least two 28-day cycles of therapy, see Appendix 10 and Appendix 8.
6. Adequate peripheral arm veins for repeated intravenous infusions
7. Life expectancy of ≥ 6 months;
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2, see Appendix 6. Patients with ECOG performance status > 2 solely based on bone pain secondary to MM may be eligible following consultation and approval of medical monitor;
9. 12-lead Electrocardiogram (ECG) with QT interval calculated by Fridericia Formula (QTcF) interval of ≤ 470 msec, see Appendix 11;
10. Adequate organ function with the following laboratory results during screening (within 21 days) and immediately before study treatment administration on Cycle 1 Day 1:

    * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm³ (1.0 x 10⁹/L) (Growth factors cannot be used within 10 days (14 days for pegfilgrastim) prior to initiation of study treatment)
    * Platelet count ≥ 75,000 cells/ mm³ (75 x 10⁹/L) (without transfusions during the 10 days prior to initiation of therapy)
    * Hemoglobin ≥ 8.0 g/dL (Red blood cell [RBC] transfusions are permitted)
    * Total Bilirubin ≤ 1.5 x upper limit of normal (ULN), except patients diagnosed with Gilbert's syndrome that have been reviewed and approved by the Medical Monitor
    * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) ≤ 3.0 x ULN
    * Renal function: Estimated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula of ≥ 45 mL/min, see Appendix 12.
11. Must have or be willing to have an acceptable central catheter (Port a Cath, peripherally inserted central catheter [PICC] line, or central venous catheter [CVC]) and a PVC;
12. a) Male patients: A male patient is eligible if he agrees to use contraception as detailed in Appendix 4 of this protocol during the treatment period and for at least 3 months after the last dose of study treatment and refrains from donating sperm during this period b) Female patients: A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: I. Not a woman of childbearing potential (WOCBP) as defined in Appendix 4 or II. A WOCBP who agrees to follow the contraceptive guidance in Appendix 4 during the treatment period and for at least 28 days after the last dose of study treatment

Exclusion Criteria:

1. Primary refractory disease (i.e. never responded with at least minimal response [MR] to any prior therapy);
2. Evidence of mucosal and/or internal bleeding or platelet transfusion refractory (platelet count fails to increase by > 10,000 cells/mm³ after a transfusion of an appropriate dose of platelets);
3. Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient or would adversely affect his/her participating in this study. Examples of such conditions are: a significant history of cardiovascular disease (e.g., myocardial infarction, significant cardiac conduction system abnormalities, uncontrolled hypertension, ≥ Grade 3 thromboembolic event in the last 6 months);
4. Known active infection that is uncontrolled or has required intravenous systemic therapy within 14 days of randomization. Patients that have required oral anti-infective treatment within 14 days of randomization should be discussed with the Medical Monitor;
5. Other malignancy diagnosed or requiring treatment within the past 3 years with the exception of adequately treated basal cell carcinoma, squamous cell skin cancer, carcinoma in-situ of the cervix or breast or very low and low risk prostate cancer in active surveillance;
6. Pregnant or breast-feeding females;
7. Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse compliance or follow-up evaluation;
8. Human immunodeficiency virus (HIV) or active hepatitis B or C viral infection;
9. Concurrent known or suspected amyloidosis or plasma cell leukemia;
10. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes);
11. Known central nervous system (CNS) or meningeal involvement of myeloma
12. Any of the following treatments, within the specified timeframe

    * Previous cytotoxic therapies, including cytotoxic investigational agents, for MM within 3 weeks (6 weeks for nitrosoureas) prior to initiation of therapy.
    * The use of live vaccines within 30 days before initiation of therapy.
    * IMiDs, PIs and or corticosteroids within 2 weeks prior to initiation of therapy.
    * Other investigational therapies and monoclonal antibodies within 4 weeks of initiation of therapy.
    * Prednisone up to but no more than 10 mg orally q.d. or its equivalent for symptom management of comorbid conditions is permitted but dose should be stable for at least 7 days prior to initiation of therapy.

    Other washout times may be considered following consultation with the medical monitor.
13. Residual side effects to previous therapy > Grade 1 prior to initiation of therapy (Alopecia any grade and/or neuropathy Grade 1 without pain are permitted);
14. Prior stem cell transplant (autologous and/or allogenic) within 6 months of initiation of therapy;
15. Prior allogeneic stem cell transplantation with active graft-versus-host-disease;
16. Prior major surgical procedure or radiation therapy within 4 weeks of the initiation of therapy (this does not include limited course of radiation used for management of bone pain within 7 days of initiation of therapy);
17. Known intolerance to the required dose and schedule of steroid therapy, as determined by the investigator;
18. Known hypersensitivity reaction to melphalan, melflufen or its excipients
19. Prior treatment with melflufen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2022-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- The Oncology Institute of Hope & Innovation - Glendale, Glendale, California, United States
- Bulgaria (2):
  - Specialized Hospital for Active Treatment of Hematological Diseases, Sofia, Sofia
  - Multiprofile Hospital for Active Treatment "Sveta Marina", Varna, Varna
- Czechia (2):
  - University Hospital Brno, Clinic of Internal Medicine - Hematology and Oncology, Brno
  - University Hospital Olomouc, Clinic of Hemato-Oncology, Olomouc
- Hungary (2):
  - Central Hospital of Southern Pest National Institute of Hematology and Infectious Diseases, Department of Hematology and Stem Cell Transplantation, Budapest
  - Semmelweis University, 3rd Department of Internal Medicine, Budapest
- Ukraine (3):
  - Public Non-Profit Enterprise "City Clinical Hospital #4" under Dnipro City Council, Regional Hematology Center, Dnipro
  - Public Non-Profit Enterprise "Kyiv City Clinical Hospital #9" under the Executive Body of Kyiv City Council, Hematology Department #1, Kyiv
  - Institute of Blood Pathology and Transfusion Medicine, Department of Hematology with Laboratory Group, Lviv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Melflufen 40 mg iv Day 1 of each 28-day cycle. Dexamethasone 40 mg po Days 1,8,15 and 22 of each 28-day cycle (20 mg for patients 75 years or older). Cycle 1 administered via a PVC and Cycle 2 and onwards melflufen administered via a CVC.
  Melflufen: Peripheral versus central administration
  Dexamethasone: Oral tablets
- Arm B: Melflufen 40 mg iv Day 1 of each 28-day cycle. Dexamethasone 40 mg po Days 1,8,15 and 22 of each 28-day cycle (20 mg for patients 75 years or older). Cycle 1 administered via a CVC and Cycle 2 administered via a PVC. From Cycle 3 and onwards melflufen administered via CVC.
  Melflufen: Peripheral versus central administration
  Dexamethasone: Oral tablets
Period: Cycle 1
Arm/Group | Arm A | Arm B
Started | 14 | 13
Discontinued | 1 | 5
Completed | 13 | 8
Not Completed | 1 | 5
Not completed — Death | 0 | 3
Not completed — Disease progression | 1 | 2
Period: Cycle 2
Arm/Group | Arm A | Arm B
Started | 13 | 8
Discontinued | 3 | 1
Completed | 10 | 7
Not Completed | 3 | 1
Not completed — Death | 0 | 1
Not completed — Disease progression | 3 | 0
Period: Cycle 3 to End of Study (EOS)
Arm/Group | Arm A | Arm B
Started | 10 | 7
Ongoing in Study at Data Cut | 0 | 0
Discontinued Study in Cycle 3 or Later | 10 | 7
Completed | 0 | 0
Not Completed | 10 | 7
Not completed — Death | 1 | 3
Not completed — Disease progression | 4 | 2
Not completed — Study terminated by Sponsor | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Customized [Count of Participants; unit: Participants]
  Age group: <65 years | 8 | 4 | 12
  Age group: >=65 - 75 years | 5 | 5 | 10
  Age group: > 75 years | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 1 | 3 | 4
  Czechia | 4 | 7 | 11
  Ukraine | 3 | 2 | 5
  Bulgaria | 6 | 1 | 7
Baseline fertility status [Count of Participants; unit: Participants] — Baseline fertility status for female participants. Population: Percentages are based on the number of female participants only.
  Participants
    number analyzed (Participants) | 7 | 7 | 14
    Potentially able to bear children | 1 | 0 | 1
    Not able to bear children | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration for Melphalan
Description: To evaluate and compare the pharmacokinetic (PK) variable Cmax of melphalan after central and peripheral intravenous infusion of melflufen.
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1. Samples were collected 5, 10, 15, 20, and 25 minutes after the start of the infusion; immediately before the end of the infusion; and 5, 10, 15, and 30 minutes and 1, 2, and 4 hours after the end of the infusion.
Population: Pharmacokinetic (PK) Set: All patients that received at least two melflufen doses of 40 mg and had sufficient PK samples taken at Cycle 1 and 2 for determination of all PK variables. One PK sampling series following peripheral administration and one PK sampling series following central administration. Patients with a dose reduction in cycle 2 were not evaluable for PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Peripheral Venous Catheter (PVC): Combined treatment ARM for all PVC administration from both ARM A & ARM B during Cycle 1 and 2. Melflufen 40 mg iv Day 1 of each 28-day cycle. Dexamethasone 40 mg po Days 1,8,15 and 22 of each 28-day cycle (20 mg for patients 75 years or older). ARM A Cycle 1 administered via a PVC and Cycle 2 and onwards melflufen administered via a CVC. ARM B Cycle 1 administered via a CVC and Cycle 2 administered via a PVC. From Cycle 3 and onwards melflufen administered via CVC. Melflufen: Peripheral versus central administration. Dexamethasone: Oral tablets.
- Central Venous Catheter (CVC): Combined treatment ARM for all CVC administration from both ARM A & ARM B during Cycle 1 and 2. Melflufen 40 mg iv Day 1 of each 28-day cycle. Dexamethasone 40 mg po Days 1,8,15 and 22 of each 28-day cycle (20 mg for patients 75 years or older). ARM A Cycle 1 administered via a PVC and Cycle 2 and onwards melflufen administered via a CVC. ARM B Cycle 1 administered via a CVC and Cycle 2 administered via a PVC. From Cycle 3 and onwards melflufen administered via CVC. Melflufen: Peripheral versus central administration. Dexamethasone: Oral tablets.
Arm/Group | Peripheral Venous Catheter (PVC) | Central Venous Catheter (CVC)
Number analyzed (Participants) | 21 | 21
ng/mL
  Cycle 1: number analyzed (Participants) | 12 | 8
  Cycle 1 | 486.1 (21.34) | 530.1 (25.23)
  Cycle 2: number analyzed (Participants) | 8 | 13
  Cycle 2 | 546.3 (31.83) | 449.2 (40.66)
Statistical Analysis 1: Comparison: Peripheral Venous Catheter (PVC) vs Central Venous Catheter (CVC); Based on a geometric mean ratio (GMR) peripheral vs. central of 0.95, a 90% confidence interval (CI) for the ratio of geometric means within bioequivalence limits of 0.8 and 1.25, and 80% power, a sample size of 20 patients (10 per sequence) was required assuming a within-patient variability for period differences (in log scale) of 0.29. Approximately 25 patients were to be enrolled to achieve 20 PK- and local tolerance-evaluable patients; Test type: Equivalence — The condition for similarity was if the 90% CI for the GMR was within the bioequivalence limits of 0.8 and 1.25; Adjusted geometric mean ratio (GMR) = 0.946, 90% CI 2-sided [0.849 to 1.053] — CVC vs. PVC, where CVC is numerator and PVC is denominator. Linear Mixed Effect Model included terms for period, sequence and administration route (PVC or CVC) as fixed effects and subject nested within sequence as a random effect

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve AUC(0-t) of Melphalan
Description: To evaluate and compare the pharmacokinetic (PK) variable AUC(0-t) of melphalan after central and peripheral intravenous infusion of melflufen.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Arm/Group | Peripheral Venous Catheter (PVC) | Central Venous Catheter (CVC)
Number analyzed (Participants) | 21 | 21
min*ng/mL
  Cycle 1: number analyzed (Participants) | 12 | 8
  Cycle 1 | 49518.36 (23.710) | 59543.20 (17.698)
  Cycle 2: number analyzed (Participants) | 8 | 13
  Cycle 2 | 60273.95 (30.037) | 46173.13 (43.336)
Statistical Analysis 1: Comparison: Peripheral Venous Catheter (PVC) vs Central Venous Catheter (CVC); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The condition for similarity was if the 90% CI for the GMR was within the bioequivalence limits of 0.8 and 1.25; Adjusted geometric mean ratio (GMR) = 0.952, 90% CI 2-sided [0.861 to 1.053] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve AUC(0-inf) of Melphalan
Description: To evaluate and compare the pharmacokinetic (PK) variable AUC(0-inf) of melphalan after central and peripheral intravenous infusion of melflufen
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Arm/Group | Peripheral Venous Catheter (PVC) | Central Venous Catheter (CVC)
Number analyzed (Participants) | 21 | 21
min*ng/mL
  Cycle 1: number analyzed (Participants) | 12 | 8
  Cycle 1 | 54216.70 (23.794) | 66835.47 (18.171)
  Cycle 2: number analyzed (Participants) | 8 | 13
  Cycle 2 | 67403.07 (30.149) | 50835.59 (44.728)
Statistical Analysis 1: Comparison: Peripheral Venous Catheter (PVC) vs Central Venous Catheter (CVC); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The condition for similarity was if the 90% CI for the GMR was within the bioequivalence limits of 0.8 and 1.25; Adjusted geometric mean ratio (GMR) = 0.955, 90% CI 2-sided [0.863 to 1.058] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Number of Participants With Local Reactions Including Phlebitis at Infusion Site After Peripheral Intravenous Administration
Description: Assessment of the local tolerability of peripheral intravenous administration of melflufen using the Visual Infusion Phlebitis (VIP) scale. The VIP scale provides a score from 0 to 5, noting an ascending order of severity of inflammation. A score of 0 is the lowest possible score, meaning no inflammation detected, and 5 is the highest score, indicating the most severe reaction.
Time Frame: 15 minutes and 4 hours after peripheral intravenous administration, pre- and post-infusion on Day 1 and Day 8
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Venous Catheter (PVC)
Number analyzed (Participants) | 27
Participants
  Cycle 1 Day 1 Pre-Infusion: number analyzed (Participants) | 13
  Cycle 1 Day 1 Pre-Infusion: VIP score = 0 | 13
  Cycle 1 Day 1 Pre-Infusion: VIP score = 1 | 0
  Cycle 1 Day 1 Pre-Infusion: VIP score = 2 | 0
  Cycle 1 Day 1 Pre-Infusion: VIP score = 3 | 0
  Cycle 1 Day 1 Pre-Infusion: VIP score = 4 | 0
  Cycle 1 Day 1 Pre-Infusion: VIP score = 5 | 0
  Cycle 1 Day 1 Post-Infusion: number analyzed (Participants) | 13
  Cycle 1 Day 1 Post-Infusion: VIP score = 0 | 13
  Cycle 1 Day 1 Post-Infusion: VIP score = 1 | 0
  Cycle 1 Day 1 Post-Infusion: VIP score = 2 | 0
  Cycle 1 Day 1 Post-Infusion: VIP score = 3 | 0
  Cycle 1 Day 1 Post-Infusion: VIP score = 4 | 0
  Cycle 1 Day 1 Post-Infusion: VIP score = 5 | 0
  Cycle 1 Day 8: number analyzed (Participants) | 10
  Cycle 1 Day 8: VIP score = 0 | 10
  Cycle 1 Day 8: VIP score = 1 | 0
  Cycle 1 Day 8: VIP score = 2 | 0
  Cycle 1 Day 8: VIP score = 3 | 0
  Cycle 1 Day 8: VIP score = 4 | 0
  Cycle 1 Day 8: VIP score = 5 | 0
  Cycle 2 Day 1 Pre-Infusion: number analyzed (Participants) | 8
  Cycle 2 Day 1 Pre-Infusion: VIP score = 0 | 8
  Cycle 2 Day 1 Pre-Infusion: VIP score = 1 | 0
  Cycle 2 Day 1 Pre-Infusion: VIP score = 2 | 0
  Cycle 2 Day 1 Pre-Infusion: VIP score = 3 | 0
  Cycle 2 Day 1 Pre-Infusion: VIP score = 4 | 0
  Cycle 2 Day 1 Pre-Infusion: VIP score = 5 | 0

5. Secondary Outcome: Peak Plasma Concentration for Melflufen and Desethyl-melflufen
Description: To evaluate and compare the pharmacokinetic (PK) variable Cmax of melflufen and desethyl-melflufen after central and peripheral intravenous infusion of melflufen.
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 - 13 PK samples during and post infusion (28 days cycle)
Population: Pharmacokinetic (PK) Analysis set: All patients that received at least two melflufen doses of 40 mg and had sufficient PK samples taken at Cycle 1 and 2 for determination of all PK variables. One PK sampling series following peripheral administration and one PK sampling series following central administration. Patients with a dose reduction in cycle 2 were not evaluable for PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Peripheral Venous Catheter (PVC) | Central Venous Catheter (CVC)
Number analyzed (Participants) | 21 | 21
ng/mL
  Melflufen Cycle 1: number analyzed (Participants) | 11 | 8
  Melflufen Cycle 1 | 151.11 (59.74) | 123.0 (47.498)
  Melflufen Cycle 2: number analyzed (Participants) | 7 | 13
  Melflufen Cycle 2 | 127.27 (75.872) | 141.75 (47.921)
  Desethyl-melflufen Cycle 1: number analyzed (Participants) | 11 | 8
  Desethyl-melflufen Cycle 1 | 16.721 (33.2618) | 11.851 (41.3587)
  Desethyl-melflufen Cycle 2: number analyzed (Participants) | 8 | 13
  Desethyl-melflufen Cycle 2 | 16.801 (43.8965) | 11.851 (41.3587)
Statistical Analysis 1: Comparison: Peripheral Venous Catheter (PVC) vs Central Venous Catheter (CVC); For melflufen: Based on a geometric mean ratio (GMR) peripheral vs central of 0.95, a 90% confidence interval (CI) for the ratio of geometric means within bioequivalence limits of 0.8 and 1.25, and 80% power, a sample size of 20 patients (10 per sequence) was required assuming a within-patient variability for period differences (in log scale) of 0.29. Approximately 25 patients were to be enrolled to achieve 20 PK- and local tolerance-evaluable patients; Test type: Equivalence — The condition for similarity was if the 90% CI for the GMR was within the bioequivalence limits of 0.8 and 1.25; adjusted geometric mean ratio (GMR) = 0.948, 90% CI 2-sided [0.736 to 1.222] — CVC vs PVC CVC is numerator and PVC is denominator. Linear Mixed Effect Model included terms for period, sequence and administration route (PVC or CVC) as fixed effects and subject nested within sequence as a random effect
Statistical Analysis 2: Comparison: Peripheral Venous Catheter (PVC) vs Central Venous Catheter (CVC); For desmethyl-melflufen: Based on a geometric mean ratio (GMR) peripheral vs central of 0.95, a 90% confidence interval (CI) for the ratio of geometric means within bioequivalence limits of 0.8 and 1.25, and 80% power, a sample size of 20 patients (10 per sequence) was required assuming a within-patient variability for period differences (in log scale) of 0.29. Approximately 25 patients were to be enrolled to achieve 20 PK- and local tolerance-evaluable patients; Test type: Equivalence — The condition for similarity was if the 90% CI for the GMR was within the bioequivalence limits of 0.8 and 1.25; [adjusted geometric mean ratio (GMR)] = 0.846, 90% CI 2-sided [0.748 to 0.957] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve AUC(0-t) of Melflufen and Desethyl-melflufen
Description: To evaluate and compare the pharmacokinetic (PK) variable AUC(0-t) of melflufen and desethyl-melflufen after central and peripheral intravenous infusion of melflufen
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 - 13 PK samples during and post infusion (28 days cycle)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min x ng/mL
Arm/Group | Peripheral Venous Catheter (PVC) | Central Venous Catheter (CVC)
Number analyzed (Participants) | 21 | 21
min x ng/mL
  Melflufen Cycle 1 (0-t): number analyzed (Participants) | 11 | 8
  Melflufen Cycle 1 (0-t) | 3617.03 (52.244) | 2828.69 (51.646)
  Melflufen Cycle 2 (0-t): number analyzed (Participants) | 7 | 13
  Melflufen Cycle 2 (0-t) | 3083.74 (80.639) | 3078.21 (49.443)
  Desethyl-melflufen Cycle 1 (0-t): number analyzed (Participants) | 11 | 8
  Desethyl-melflufen Cycle 1 (0-t) | 563.34 (42.086) | 639.39 (34.053)
  Desethyl-melflufen Cycle 2 (0-t): number analyzed (Participants) | 8 | 13
  Desethyl-melflufen Cycle 2 (0-t) | 636.06 (51.627) | 391.11 (49.458)
Statistical Analysis 1: Comparison: Peripheral Venous Catheter (PVC) vs Central Venous Catheter (CVC); Based on a geometric mean ratio (GMR) peripheral vs central of 0.95, a 90% confidence interval (CI) for the ratio of geometric means within bioequivalence limits of 0.8 and 1.25, and 80% power, a sample size of 20 patients (10 per sequence) was required assuming a within-patient variability for period differences (in log scale) of 0.29. Approximately 25 patients were to be enrolled to achieve 20 PK- and local tolerance-evaluable patients; Test type: Equivalence — The condition for similarity was if the 90% CI for the GMR was within the bioequivalence limits of 0.8 and 1.25; adjusted geometric mean ratio (GMR) = 0.877, 90% CI 2-sided [0.684 to 1.126] — Data above refer to meflufen. CVC vs PVC CVC is numerator, PVC is denominator. Linear Mixed Effect Model included terms for period, sequence and administration route (PVC or CVC) as fixed effects and subject nested within sequence as a random effect
Statistical Analysis 2: Comparison: Peripheral Venous Catheter (PVC) vs Central Venous Catheter (CVC); [analysis description as in outcome 6, analysis 1]; Test type: Equivalence — The condition for similarity was if the 90% CI for the GMR was within the bioequivalence limits of 0.8 and 1.25; adjusted geometric mean ratio (GMR) = 0.897, 90% CI 2-sided [0.819 to 0.982] — Data above refer to desethyl-melflufen. CVC vs PVC CVC is numerator, PVC is denominator. Linear Mixed Effect Model included terms for period, sequence and administration route as fixed effects and subject nested within sequence as a random effect

7. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve AUC(0-inf) of Melflufen and Desethyl-melflufen
Description: To evaluate and compare the pharmacokinetic (PK) variable AUC(0-inf) of melflufen and desethyl-melflufen after central and peripheral intravenous infusion of melflufen
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 - 13 PK samples during and post infusion (28 days cycle)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min x ng/mL
Arm/Group | Peripheral Venous Catheter (PVC) | Central Venous Catheter (CVC)
Number analyzed (Participants) | 21 | 21
min x ng/mL
  Melflufen Cycle 1 (0-inf): number analyzed (Participants) | 11 | 8
  Melflufen Cycle 1 (0-inf) | 3639.34 (52.379) | 2841.23 (51.631)
  Meflufen Cycle 2 (0-inf): number analyzed (Participants) | 7 | 13
  Meflufen Cycle 2 (0-inf) | 3099.70 (80.708) | 3093.96 (49.295)
  Desethyl-melflufen Cycle 1 (0-inf): number analyzed (Participants) | 11 | 8
  Desethyl-melflufen Cycle 1 (0-inf) | 609.44 (40.778) | 759.25 (34.619)
  Desethyl-melflufen Cycle 2 (0-inf): number analyzed (Participants) | 8 | 13
  Desethyl-melflufen Cycle 2 (0-inf) | 695.29 (51.722) | 440.65 (43.547)
Statistical Analysis 1: Comparison: Peripheral Venous Catheter (PVC) vs Central Venous Catheter (CVC); [analysis description as in outcome 6, analysis 1]; Test type: Equivalence — The condition for similarity was if the 90% CI for the GMR was within the bioequivalence limits of 0.8 and 1.25; adjusted geometric mean ratio (GMR) = 0.877, 90% CI 2-sided [0.684 to 1.124] — Data above refer to melflufen. CVC vs PVC CVC is numerator, PVC is denominator. Linear Mixed Effect Model included terms for period, sequence & administration route (PVC or CVC) as fixed effects and subject nested within sequence as a random effect
Statistical Analysis 2: Comparison: Peripheral Venous Catheter (PVC) vs Central Venous Catheter (CVC); [analysis description as in outcome 6, analysis 1]; Test type: Equivalence — The condition for similarity was if the 90% CI for the GMR was within the bioequivalence limits of 0.8 and 1.25; adjusted geometric mean ratio (GMR) = 0.908, 90% CI 2-sided [0.833 to 0.989] — Data above refer to desethyl-melflufen. CVC vs PVC CVC is numerator, PVC is denominator. Linear Mixed Effect Model included terms for period, sequence & administration route as fixed effects and subject nested within sequence as a random effect

8. Secondary Outcome: Elimination Half-life (t1/2) of Melflufen, Melphalan and Desethyl-melflufen
Description: To evaluate elimination half-life (t½) for melflufen, melphalan and desethyl-melflufen after central and peripheral intravenous infusion of melflufen.
Time Frame: Cycle 1 Day 1 and Cycle 2 Day 1 - 13 measurements during and post infusion (28 days cycle)
Population: Pharmacokinetic (PK) Analysis set:All patients that received at least two melflufen doses of 40 mg and had sufficient PK samples taken at Cycle 1 and 2 for determination of all PK variables. One PK sampling series following peripheral administration and one PK sampling series following central administration. Patients with a dose reduction in cycle 2 were not evaluable for PK.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Peripheral Venous Catheter (PVC) | Central Venous Catheter (CVC)
Number analyzed (Participants) | 21 | 21
minutes
  Melphalan Cycle 1: number analyzed (Participants) | 12 | 8
  Melphalan Cycle 1 | 72.51 (14.993) | 80.09 (12.85)
  Melphalan Cycle 2: number analyzed (Participants) | 8 | 13
  Melphalan Cycle 2 | 78.09 (18.118) | 72.97 (16.84)
  Melflufen Cycle 1: number analyzed (Participants) | 11 | 8
  Melflufen Cycle 1 | 7.42 (106.832) | 4.45 (90.634)
  Melflufen Cycle 2: number analyzed (Participants) | 7 | 13
  Melflufen Cycle 2 | 6.15 (81.278) | 5.74 (80.837)
  Desethyl-melflufen Cycle 1: number analyzed (Participants) | 11 | 8
  Desethyl-melflufen Cycle 1 | 18.44 (49.68) | 23.49 (43.423)
  Desethyl-melflufen Cycle 2: number analyzed (Participants) | 8 | 13
  Desethyl-melflufen Cycle 2 | 25.04 (83.298) | 17.43 (37.708)

9. Secondary Outcome: Frequency of Treatment-Emergent Adverse Events (TEAEs) by MedDRA SOC and PT
Description: To assess safety and general tolerability of melflufen by collecting non-serious Adverse Events (AEs) from the start of study treatment until 30 days after the last dose of any study drug (melflufen or dexamethasone) or initiation of subsequent therapy whichever occurred first. Serious AEs (SAEs) were collected from the time the subject signed the ICF until 30 days after the last dose of any study drug (melflufen or dexamethasone) or initiation of subsequent therapy whichever occurred first.
Time Frame: Median treatment durations for Arm A and Arm B were 29.14 weeks and 12.14 weeks, respectively. The AE reporting period is estimated to be 30 days longer.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Arm A plus Arm B
Arm/Group | Arm A | Arm B | Overall
Number analyzed (Participants) | 14 | 13 | 27
Participants
  Patients with at least 1 TEAE | 13 | 13 | 26
  Blood and lymphatic system disorders | 13 | 12 | 25
  Thrombocytopenia | 10 | 10 | 20
  Neutropenia | 9 | 9 | 18
  Anaemia | 9 | 7 | 16
  Leukopenia | 2 | 1 | 3
  Infections and Infestations | 6 | 7 | 13
  Pneumonia | 3 | 2 | 5
  COVID-19 pneumonia | 0 | 3 | 3
  Respiratory tract infection | 2 | 0 | 2
  General disorders and administration site conditions | 5 | 6 | 11
  Pyrexia | 2 | 3 | 5
  Fatigue | 1 | 2 | 3
  General health deterioration | 0 | 2 | 2
  Musculoskeletal and connective tissue disorders | 4 | 5 | 9
  Arthralgia | 1 | 2 | 3
  Back pain | 2 | 1 | 3
  Bone pain | 2 | 0 | 2
  Investigations | 4 | 4 | 8
  SARS-CoV-2 test positive | 2 | 4 | 6
  C-reactive protein increased | 2 | 0 | 2
  Injury, poisoning and procedural complications | 0 | 3 | 3
  femur fracture | 0 | 2 | 2
  Skin and subcutaneous tissue disorders | 2 | 0 | 2
  Rash | 2 | 0 | 2

10. Secondary Outcome: Best Response (Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), Minimal Response (MR), Stable Disease (SD) or Progressive Disease (PD)
Description: To assess best response during the study with the criteria established by the International Myeloma Working Group Uniform Response Criteria (IMWG-URC) for sCR, CR, VGPR, PR, SD and PD
Time Frame: From initiation of therapy until disease progression. Median treatment durations for Arm A and Arm B were 29.14 weeks and 12.14 weeks, respectively.
Population: Full Analysis Set: 14 participants randomized to Arm A and 13 participants randomized to Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Overall
Number analyzed (Participants) | 14 | 13 | 27
Participants
  Stringent complete response | 0 | 0 | 0
  Complete response | 1 | 0 | 1
  Very good partial response | 0 | 0 | 0
  Partial response | 3 | 1 | 4
  Minimal response | 4 | 1 | 5
  Stable disease | 2 | 6 | 8
  Progressive disease | 2 | 1 | 3
  Not available | 2 | 4 | 6

11. Secondary Outcome: ORR
Description: To assess overall response rate (ORR), including CR/sCR, VGPR and PR, during the study with the criteria established by the IMWG-URC.
Time Frame: From initiation of therapy until disease progression. Maximum treatment durations for Arm A and Arm B were 68.4 and 59.0 weeks, respectively.
Population: Full Analysis set: 14 participants randomized to Arm A and 13 participants randomized to Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Overall
Number analyzed (Participants) | 14 | 13 | 27
Participants | 4 | 1 | 5

12. Secondary Outcome: CBR
Description: To assess clinical benefit rate (CBR), i.e., proportion of patients that achieve a confirmed minimal response or better (sCR, CR, VGPR, PR and MR), during the study with the criteria established by the IMWG-URC.
Time Frame: To be assessed at the end of study drug treatment. Maximum treatment durations for Arm A and Arm B were 68.4 and 59.0 weeks, respectively.
Population: Full Analysis set: 14 participants randomized to Arm A and 13 participants randomized to Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Overall
Number analyzed (Participants) | 14 | 13 | 27
Participants | 8 | 2 | 10

13. Secondary Outcome: DOR
Description: To assess duration of response (DOR): the time in months from the first evidence of confirmed assessment of sCR, CR, VGPR, or PR to first confirmed disease progression according to the criteria established by the IMWG-URC or to death due to any cause. DOR is defined only for patients with a confirmed PR or better.
Time Frame: From confirmed response until disease progression. Maximum treatment durations for Arm A and Arm B were 68.4 and 59.0 weeks, respectively.
Population: Full Analysis set: 14 participants randomized to Arm A and 13 participants randomized to Arm B.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B | Overall
Number analyzed (Participants) | 14 | 13 | 27
months | NA [1.18 to NA] — Note: At study termination, the DOR data was insufficient to evaluate due to the low number of patient events: 1 (7.1%) in Arm A, 0 in Arm B. | NA [NA to NA] — Note: At study termination, the DOR data was insufficient to evaluate due to the low number of patient events: 1 (7.1%) in Arm A, 0 in Arm B. | NA [1.18 to NA] — Note: At study termination, the DOR data was insufficient to evaluate due to the low number of patient events: 1 (7.1%) in Arm A, 0 in Arm B.

14. Secondary Outcome: DOCB
Description: To assess duration of clinical benefit (DOCB) in patients with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), PR, or MR during the study with the criteria established by the IMWG-URC.
Time Frame: From first evidence of confirmed assessment of sCR, CR, VGPR, PR or MR to first confirmed disease progression, or to death due to any cause. Maximum treatment durations for Arm A and Arm B were 68.4 and 59.0 weeks, respectively.
Population: Full Analysis set: 14 participants randomized to Arm A and 13 participants randomized to Arm B.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B | Overall
Number analyzed (Participants) | 14 | 13 | 27
months | NA [3.02 to NA] — Overall, 3 patients had experienced an event and 7 had been censored, as they were alive and without a PD assessment at the time of study termination. Consequently, the DOCB data was insufficient to evaluate. | NA [NA to NA] — Overall, 3 patients had experienced an event and 7 had been censored, as they were alive and without a PD assessment at the time of study termination. Consequently, the DOCB data was insufficient to evaluate. | NA [7.16 to NA] — Overall, 3 patients had experienced an event and 7 had been censored, as they were alive and without a PD assessment at the time of study termination. Consequently, the DOCB data was insufficient to evaluate.

15. Secondary Outcome: TTR
Description: To assess time to response (TTR) in patients with PR or better during the study with the criteria established by the UMWG-URC.
Time Frame: From initiation of therapy until documented disease response. Maximum treatment durations for Arm A and Arm B were 68.4 and 59.0 weeks, respectively.
Population: Full Analysis set:14 participants randomized to Arm A and 13 participants randomized to Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Overall
Number analyzed (Participants) | 14 | 13 | 27
Participants | 4 | 1 | 5

16. Secondary Outcome: TTP
Description: To assess time to progression (TTP) during the study with the criteria established by the IMWG-URC.
Time Frame: From date of randomization until documented disease progression. Maximum treatment durations for Arm A and Arm B were 68.4 and 59.0 weeks, respectively.
Population: Full Analysis set: 14 participants randomized to Arm A and 13 participants randomized to Arm B.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B | Overall
Number analyzed (Participants) | 14 | 13 | 27
months | 5.78 [2.73 to NA] — Overall, 13 (48.1%) patients had experienced progression and 14 (51.9%) were censored, as they were alive and lacked PD assessments or documentation at the time of study termination | 4.80 [2.79 to NA] — Overall, 13 (48.1%) patients had experienced progression and 14 (51.9%) were censored, as they were alive and lacked PD assessments or documentation at the time of study termination | 5.78 [3.06 to NA] — Overall, 13 (48.1%) patients had experienced progression and 14 (51.9%) were censored, as they were alive and lacked PD assessments or documentation at the time of study termination

17. Secondary Outcome: TTNT
Description: To assess time to next treatment (TTNT)
Time Frame: From randomization to the date of next anti-myeloma treatment. Maximum treatment durations for Arm A and Arm B were 68.4 and 59.0 weeks, respectively.
Population: Full Analysis set: 14 participants randomized to Arm A and 13 participants randomized to Arm B.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B | Overall
Number analyzed (Participants) | 14 | 13 | 27
months | NA [NA to NA] — In this study, patients were followed to progression. No patients had a new treatment for MM prior to progression, and as a result TTNT was not calculable. | NA [NA to NA] — In this study, patients were followed to progression. No patients had a new treatment for MM prior to progression, and as a result TTNT was not calculable. | NA [NA to NA] — In this study, patients were followed to progression. No patients had a new treatment for MM prior to progression, and as a result TTNT was not calculable.

18. Secondary Outcome: PFS
Description: To assess progression free survival (PFS)
Time Frame: From initiation of therapy until documented disease progression or initiation of new therapy. Maximum treatment durations for Arm A and Arm B were 68.4 and 59.0 weeks, respectively.
Population: Full Analysis set: 14 participants randomized to Arm A and 13 participants randomized to Arm B.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B | Overall
Number analyzed (Participants) | 14 | 13 | 27
months | 5.21 [2.73 to NA] — Overall, 19 (70.4%) patients experienced progression during the study and 8 (29.6%) were censored, due to lack of PD assessments or deaths at the time of study termination. | 2.89 [1.51 to 4.60] | 3.73 [2.73 to 5.78]

19. Secondary Outcome: Grade 3/4 Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 9
Time Frame: Median treatment durations for Arm A and Arm B were 29.14 and 12.14 weeks, respectively. The AE reporting period is estimated to be 30 days longer.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Grade 3/4: Melflufen 40 mg IV Day 1 of each 28 day cycle. Dexamethasone 40 mg PO Days 1, 8, 15 and 22 of each 28 day cycle; if >75 yr of age 20 mg. Cycle 1will be administered via peripheral venous catheter (PVC) and Cycle 2 onwards melflufen will be administered via a central venous catheter (CVC).
  Melphalan: PVC vs CVC administration Dexamethasone: oral tablets
- Arm B: Grade 3/4: Melflufen 40 mg IV Day 1 of each 28 day cycle. Dexamethasone 40 mg PO Days 1, 8, 15 and 22 of each 28 day cycle; if >75 yr of age 20 mg. Cycle 1 will be administered via central venous catheter (CVC). Cycle 2 will be administered via peripheral venous catheter (PVC). From Cycle 3 and onwards melflufen will be administered via CVC.
  Melphalan: PVC vs CVC administration Dexamethasone: oral tablets
- Overall: Grade 3/4: Arm A plus Arm B
Arm/Group | Arm A: Grade 3/4 | Arm B: Grade 3/4 | Overall: Grade 3/4
Number analyzed (Participants) | 14 | 13 | 27
Participants
  Blood and lymphatic system disorders | 12 | 10 | 22
  Thrombocytopenia | 8 | 10 | 18
  Neutropenia | 8 | 7 | 15
  Anaemia | 5 | 3 | 8
  Leukopenia | 2 | 1 | 3
  Lymphopenia | 1 | 1 | 2
  Febrile neutropenia | 1 | 1 | 2
  Infections and infestations | 2 | 2 | 4
  Pneumonia | 2 | 1 | 3
  COVID-19 pneumonia | 0 | 1 | 1
  Sepsis | 1 | 0 | 1
  General disorders and administration site conditions | 0 | 0 | 0
  General physical health deterioration | 0 | 0 | 0
  Death | 0 | 0 | 0
  Asthenia | 0 | 1 | 1
  Injury, poisoning and procedural complications | 0 | 3 | 3
  Femur fracture | 0 | 2 | 2
  Femoral neck fracture | 0 | 1 | 1
  Gastrointestinal disorders | 0 | 1 | 1
  Stomatitis | 0 | 1 | 1
  Musculoskeletal and connective tissue disorders | 1 | 1 | 2
  Back pain | 1 | 0 | 1
  Musculoskeletal chest pain | 0 | 1 | 1
  Nervous system disorders | 1 | 0 | 1
  Ischaemic stroke | 1 | 0 | 1
  Vascular disorders | 0 | 1 | 1
  Hypertension | 0 | 1 | 1

20. Secondary Outcome: Grade 5 Treatment-Emergent Adverse Events (TEAEs)
Description: To assess safety and general tolerability of melflufen by collecting serious adverse events (SAEs) from the signing of the ICF until 30 days after the last dose of any study drug (melflufen or dexamethasone) or initiation of subsequent therapy whichever comes first.
Time Frame: From signing of the ICF until 30 days after the last dose of any study drug or initiation of subsequent therapy, whichever comes first. Median treatment durations for Arms A and B were 29.14 weeks and 12.14 weeks. AE reporting period=30 days longer
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Grade 5: Melflufen 40 mg IV Day 1 of each 28 day cycle. Dexamethasone 40 mg PO Days 1, 8, 15 and 22 of each 28 day cycle; if >75 yr of age 20 mg. Cycle 1will be administered via peripheral venous catheter (PVC) and Cycle 2 onwards melflufen will be administered via a central venous catheter (CVC).
  Melphalan: PVC vs CVC administration Dexamethasone: oral tablets
- Arm B: Grade 5: Melflufen 40 mg IV Day 1 of each 28 day cycle. Dexamethasone 40 mg PO Days 1, 8, 15 and 22 of each 28 day cycle; if >75 yr of age 20 mg. Cycle 1 will be administered via central venous catheter (CVC). Cycle 2 will be administered via peripheral venous catheter (PVC). From Cycle 3 and onwards melflufen will be administered via CVC.
  Melphalan: PVC vs CVC administration Dexamethasone: oral tablets
- Overall: Grade 5: Arm A plus Arm B
Arm/Group | Arm A: Grade 5 | Arm B: Grade 5 | Overall: Grade 5
Number analyzed (Participants) | 14 | 13 | 27
Participants
  Infections and infestations | 0 | 3 | 3
  Pneumonia | 0 | 1 | 1
  COVID-19 pneumonia | 0 | 2 | 2
  General disorders and administration site conditions | 0 | 3 | 3
  General physical health deterioration | 0 | 2 | 2
  Death | 0 | 1 | 1
  Gastrointestinal disorders | 1 | 0 | 1
  Ileus | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: SAEs were collected from signing of the ICF until 30 days after last dose of study treatment or initiation of subsequent therapy, whichever occurred first. Non-serious AEs were collected from the start of study treatment until 30 days after the last dose of any study drug or initiation of subsequent therapy, whichever occurred first. Median treatment durations for Arm A and Arm B were 29.14 weeks and 12.14 weeks, respectively. The AE reporting period is estimated to be 30 days longer.
Description: Adverse events cannot be compared for Arm A versus Arm B. Because of the crossover design of the study, all patients had a different route of administration in Cycle 2 than Cycle 1, and later AEs could be due to a cumulative effect of multiple treatment cycles. Thus, AEs occurring in Cycle 2 and beyond cannot be attributed to only 1 route of administration.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 1/14 | 8/13
Serious Adverse Events (participants affected / at risk) | 5/14 | 9/13
Other Adverse Events (participants affected / at risk) | 13/14 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=14) | Arm B (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 2 (2)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 3 (4)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=14) | Arm B (N=13)
Anaemia (Blood and lymphatic system disorders) | 9 (16) | 7 (12)
Leukopenia (Blood and lymphatic system disorders) | 2 (7) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 9 (36) | 9 (33)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (34) | 10 (23)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (2) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (3)
COVID-19 (Infections and infestations) | 1 (1) | 1 (2)
Infection (Infections and infestations) | 1 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 2 (3) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 2 (2) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Vascular pain (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT04412707/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT04412707/SAP_001.pdf